CLINICAL TRIAL: NCT03160638
Title: A Prospective, Randomized Pilot Study of the Immunomodulatory Effects of Azithromycin in Adults With Pulmonary Tuberculosis
Brief Title: Azithromycin as Host-directed Therapy for Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, Principal Investigator, PharmD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZT_DSTB_BB
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Azithromycin; Immunomodulation; Pharmacokinetics; Tissue degradation; Tissue remodelling
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin arm (Experimental): Patients in this arm will be treated with azithromycin 250 mg once daily on top of standard HRZE treatment.
  Interventions: Drug: Azithromycin 250 mg
- Standard of care arm (No Intervention): Patients in this arm will receive no additional treatment on top of standard HRZE treatment

INTERVENTIONS:
Drug: Azithromycin 250 mg — Patients will be treated with azithromycin 250 mg once daily for 28 days. An azithromycin loading dose of 500 mg (two tablets of 250 mg) will be administered on day 1
  Arms: Azithromycin arm

SUMMARY:
Rationale:

Treatment in tuberculosis (TB) is focused on eradication of the bacterial infection, however, after treatment approximately half of patients are left with a significant and permanent respiratory impairment. Adjunctive host-directed therapies are being investigated to modulate host immune responses to target mycobacterium tuberculosis (Mtb) infection and/or reduce excessive inflammation, prevent pathological tissue damage, preserve lung function and enhance effectiveness of standard drug therapy, while nonetheless eliminating Mtb. Macrolide antibiotics have previously been used in the treatment of multidrug-resistant TB. In addition to their antibiotic effects, macrolides have also been recognized to induce anti-inflammatory and immunomodulatory effects in other lung diseases.

Objective:

To investigate the immunomodulatory effects of azithromycin in tuberculosis patients receiving standard therapy (isoniazid, rifampicin, pyrazinamide, ethambutol (HRZE))

Study design:

A prospective, randomized open label intervention trial to investigate the immunomodulatory effects of azithromycin

Study population: 24

Intervention: azithromycin 250 mg once daily or standard of care (control)

Main study parameters/endpoints:

1. To assess whether azithromycin enhances resolution of systemic inflammation in patients with drug susceptible pulmonary TB receiving standard treatment.
2. To assess whether azithromycin on top of standard treatment in patients with drug susceptible pulmonary TB reduces airway inflammation and reduces tissue degradation and remodeling
3. To investigate whether these effects are associated within shortening of the time to sputum conversion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of drug sensitive pulmonary tuberculosis (molecular test; identification Mtb complex; absence of resistance genes such as rpob, inha, katg)
* Written informed consent

Exclusion Criteria:

* Patient reported previous history of treatment for tuberculosis
* Patients younger than 18 years
* Pregnancy or breast feeding
* Patients with hypersensitivity to macrolide antibiotics
* Treatment with any macrolide in the previous month
* Treatment with any tetracycline in the previous month
* Treatment with any inhaled or oral corticosteroid in the previous month
* Concomitant treatment with analgesic (NSAIDs)/immunosuppressant drugs (except paracetamol).
* Treatment with digoxin
* Patients with gastrointestinal complaints, like diarrhea and vomiting (≥grade 2, observed)
* Other known respiratory diseases, including bronchiectasis, pulmonary fibrosis, pulmonary vascular disease or lung cancer
* HIV-1 infection or AIDS
* Impaired liver function (Child-Pugh score C)
* Patients with a known QTc ≥500 ms. An electrocardiogram (ECG) will be recorded.
* Inability to spontaneously produce sputum upon diagnosis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Systemic inflammation | Before randomization, day 7 and day 28
  Changes in total & differential white blood cell counts markers
Systemic inflammation | Before randomization, day 7 and day 28
  Changes in serum inflammatory markers

SECONDARY OUTCOMES:
Pulmonary inflammation | Before randomization and day 28
  Changes in total and differential sputum inflammatory cell counts
Pulmonary inflammation | Before randomization and day 28
  Changes in cytokine levels in sputum
Pulmonary tissue degradation | Before randomization and day 28
  Changes in markers of tissue degradation in sputum
Pulmonary tissue degradation | Before randomization, day 7 and day 28
  Changes in markers of tissue degradation in serum
Pulmonary tissue remodeling | Before randomization and day 28
  Changes in markers of tissue remodeling in sputum
Pulmonary tissue remodeling | Before randomization, day 7 and day 28
  Changes in markers of tissue remodeling in serum

OTHER OUTCOMES:
Evaluation of HRZE treatment outcomes | Up to 6 months
  Time to sputum conversion
Evaluation of HRZE treatment outcomes | Up to 6 months
  Drug exposure of HRZE in relation to minimal inhibitory concentration (MIC) of Mtb for HRZE
Drug exposure of azithromycin | Day 7
  AUC0-24h of azithromycin in TB
Drug exposure of azithromycin | Day 7
  Metabolic clearance (CLm) of azithromycin in TB
Drug exposure of azithromycin | Day 7
  Volume of distribution (V) of azithromycin in TB
Drug exposure of azithromycin | Day 7
  Elimination half-life (T1/2) of azithromycin in TB

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dekkers BGJ, Kerstjens HAM, Breisnes HW, Leeming DJ, Anthony RM, Frijlink HW, van der Werf TS, Kosterink JGW, Alffenaar JC, Akkerman OW. Azithromycin as Host-Directed Therapy for Pulmonary Tuberculosis: A Randomized Pilot Trial. J Infect Dis. 2025 Jun 2;231(5):e891-e900. doi: 10.1093/infdis/jiaf069. PMID 39932906